CLINICAL TRIAL: NCT04054960
Title: A Trial of tPCS on Parkinson's Disease OFF State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114200
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease OFF state, Noninvasive stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real tPCS (Experimental): Patients will be randomized to any of the 3 arms. In Real tPCS arm, we will give active tPCS for 20 mins.
  Interventions: Device: Active tPCS
- Sham tPCS (Sham Comparator): Patients will be randomized to any of the 3 arms. In Sham tPCS arm, we will give sham tPCS for 20 mins.
  Interventions: Device: Sham tPCS
- Levodopa (Active Comparator): Patients will be randomized to any of the 3 arms. In Levodopa arm, we will give 3 tablets of Levodopa-Carbidopa (100/25).
  Interventions: Drug: Levodopa tablet

INTERVENTIONS:
Device: Active tPCS — Active anodal tPCS will be given for 20 mins to motor cortex (M1) or supplementary motor area (SMA), based on our quantitative EEG findings.
  Arms: Real tPCS
Device: Sham tPCS — For the sham condition, the electrode placement will be the same, but the electric current will be ramped down 5 seconds after the beginning of the stimulation.
  Arms: Sham tPCS
Drug: Levodopa tablet — We will give 3 tablets of Levodopa-Carbidopa (100/25).
  Arms: Levodopa

SUMMARY:
A significant number of patients with Parkinson's disease (PD) face motor fluctuations even after repeated titration of the dosing of Levodopa. Dealing with OFF state really becomes problematic for them. Aggravation of bradykinesia, rigidity, tremor and gait difficulty are the common problems in OFF state. Studies are going on drugs like Apomorphine as rescue therapy in OFF state. Recently there are studies with Noninvasive brain stimulation, as an evolving therapeutic option in different neurodegenerative diseases. In this study, the investigators are to evaluate the efficacy of transcranial pulsed current stimulation (tPCS) in the OFF state in PD patients. The investigators will give stimulation via tPCS (active/sham). EEG, Kinematic measurement of upper limb movement via KinArm, Unified Parkinson's Disease Rating Scale (UPDRS) scoring will be done and gait will be assessed via Gait Carpet - pre and post-stimulation. The investigators will evaluate the effectiveness of tPCS as a single modality or in combination with Levodopa in managing OFF state of PD.

DETAILED DESCRIPTION:
This will be a randomized sham-controlled trial. The investigators have planned to study the efficacy of Transcranial pulsed current stimulation (tPCS) in patients of Parkinson's disease (PD) in their OFF state. Each patient will come in 3 separate days in OFF state. They will first receive either active tPCS or sham tPCS or 3 tabs of Levodopa (100/25) in OFF state. Pre and post intervention analysis will be done. In those, who are receiving tPCS (active/sham), the investigators will give them Levodopa (100/25) after post stimulation assessment done. The patients will be assessed clinically by UPDRS III. EEG (for electrophysiological analysis), Gait Carpet (for Gait analysis) will also be done - before and after a single session of 20 min stimulation via tPCS. The investigators will also compare the effect of tPCS in OFF state, with that of Levodopa in OFF state.

The assessment will be done by-

1. Unified Parkinson's disease rating scale III (UPDRS III)
2. Gait via Gait Carpet
3. Quantitative Electroencephalography (qEEG)
4. KinARM

Transcranial pulsed current stimulation (tPCS) will be delivered through a pair of saline-soaked (0.9% NaCl) surface sponge electrodes. For this experiment, 20 minutes of stimulation will be performed. The stimulation would be done to the motor cortex (M1) or supplementary motor area (SMA), based on quantitative electroencephalography (qEEG) findings. For the sham stimulation, the electrode placement will be same, but the electric current will be ramped down 5 seconds.

Zeno Walkway is a pressure sensitive electronic roll-up walkway that measures the temporal and spatial parameters of gait which could in turn help in identifying any abnormalities in the gait. The patient walks on the Zeno Walkway mat before and after the tPCS stimulation to find the difference in the gait motion. The Zeno walkway will be used in conjunction with the ProtoKinetics Movement Analysis Software (PKMAS). These data will be captured and collated via the PKMAS software, resulting in numerous spatial, temporal and pressure-related gait parameters. Timed-up-and-go (TUG) (1-5minutes per trial) will be performed. The test consists of rising from chair, walking across the 20-foot gait carpet, turning around off the carpet, walking back and sitting down. This will be performed over 3 trials. Gait analysis provides various additional parameters as output such as stride length, line of progression, step length, toe-offs and other temporal and spatial parameters for analysis.

Quantitative EEG signals will be recorded, eyes-closed, no-task, using g.Nautilus g.tec wireless system. The g.tech system uses earclip reference sensors. The patient will be in a quiet place with less light or electromagnetic perturbations. During the resting state recordings, patients are seated in a comfortable arm chair and will be instructed to keep relaxed, with their eyes closed for 5 min.

Kinarm will be used to measure the kinematics of upper limb movements, via Reaching tasks. This is basically mechanical handle driven by multiple actuators. A software named BKIN will be used to setup this hardware. The Kinarm initially provides the patients with multiple points to reach in the screen and the patients would try to reach these points using the kinarm handle. The motion of the patients when trying to reach for these points is analysed by kinarm and the data would be provided to us based on this analysis.

An paired t test will be used to compare baseline data and post tPCS data. Descriptive analysis of the neurological examination findings will be provided. The output from the KinARM, gait carpet, EEG will be used for further analysis to build a descriptive machine learning model.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Idiopathic Parkinson's disease (IPD).

Exclusion Criteria:

* Parkinson plus syndromes.
* Drug-induced parkinsonism.
* Patients who cannot walk independently or wheelchair-bound.
* Patients who are not able to provide informed consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in Unified Parkinson's disease rating scale (UPDRS) part III | 3 months
  The effectiveness of tPCS in OFF state of PD will be evaluated. Unified Parkinson's disease rating scale (UPDRS) part III will be applied - pre and post stimulation. UPDRS Part III is motor examination that consists of speech, facial expression, rigidity, rest tremor, postural/action tremor, rapid alternating movements for testing bradykinesia, arising from chair, posture, gait, body bradykinesia, postural stability. In each subset, minimum score is 0 and maximum is 4. By adding, total UPDRS part III score is minimum 0 to maximum 108. Higher score means more severity of parkinsonism.
Changes in spatiotemporal gait measures using objective gait analysis | 3 months
  Zeno Walkway Gait carpet will be used and the spatiotemporal details of the gait will be analyzed by ProtoKinetics Movement Analysis Software (PKMAS) software, pre and post stimulation.
Change in upper limb motor kinetics | 3 months
  KinArm will be used pre and post stimulation to have objective measurement of upper limb motor function. Reaching task will be performed using standardized KinArm protocol. Visuomotor function of upper limb will be analyzed by postural control of arm with respect to x and y co-ordinates, angular velocity, acceleration, force and torque.
Changes in Network fragmentation using Quantitative Electroencephalography (EEG) | 3 months
  Network fragmentation will be analyzed by 5 mins of resting quantitative Electroencephalography (EEG), pre and post stimulation. All frequency bands will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alon G, Yungher DA, Shulman LM, Rogers MW. Safety and immediate effect of noninvasive transcranial pulsed current stimulation on gait and balance in Parkinson disease. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1089-95. doi: 10.1177/1545968312448233. Epub 2012 May 10. PMID 22581566